CLINICAL TRIAL: NCT06916338
Title: Clinical Study of 18F-Labeled FAPI-04 in PET Imaging of Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Weifang People's Hospital (Other); Zibo Central Hospital (Other Government); Qianfoshan Hospital (Other); Jining Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: QDFY-NM-25001
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-FAPI-04 PET scan
  Interventions: Radiation: 18F-FAPI-04 PET scan

INTERVENTIONS:
Radiation: 18F-FAPI-04 PET scan — FAPI-04, labeled with PET radio-nuclide 18F will be used as a molecular imaging tracer for PET scan. All participants will undergo 18F-FAPI-04 PET scan.

SUMMARY:
This study aims to evaluate the diagnostic accuracy (sensitivity, specificity, positive/negative predictive value, and overall accuracy) of 18F-FAPI-04 PET imaging in breast cancer for detecting fibroblast activation protein (FAP)-rich lesions. Additionally, the study will longitudinally monitor dynamic changes in FAP expression levels and tumor size during therapy, including chemotherapy, targeted therapy, or immunotherapy.The non-invasive nature of 18F-FAPI-04 PET addresses limitations of traditional biopsy-dependent stromal evaluation, offering whole-body quantification of tumor microenvironment dynamics to optimize therapeutic decision-making.

DETAILED DESCRIPTION:
Breast cancer diagnosis and treatment continue to face challenges in adequately assessing tumor heterogeneity and dynamically monitoring therapeutic responses. Traditional biopsy-dependent pathological analysis is limited by its invasive nature, sampling bias, and inability to repeatedly sample tissues, making it difficult to capture the spatiotemporal heterogeneity of cancer-associated fibroblasts (CAFs) within the systemic tumor microenvironment (TME). Fibroblast activation protein (FAP), a core marker of CAFs, plays a critical role in tumor proliferation, metastasis, immune evasion, and drug resistance, with its expression levels significantly correlating with patient prognosis. However, current imaging techniques, such as 18F-FDG PET, primarily reflect tumor metabolic activity and lack sufficient sensitivity for detecting FAP-positive lesions with low metabolism but high aggressiveness. They also fail to differentiate post-therapy inflammatory responses from residual tumor activity. 18F-FAPI-04 PET overcomes these biological limitations of conventional imaging by precisely targeting FAP, enabling non-invasive molecular visualization of systemic lesions. Its high target-to-background ratio allows detection of early-stage micrometastases (e.g., lymph node or bone metastases), addressing the risk of missed diagnoses with FDG PET. Furthermore, by quantifying dynamic changes in FAP expression, it enables real-time monitoring of therapy-induced stromal remodeling (e.g., CAF depletion post-immunotherapy or pro-fibrotic responses post-chemotherapy), providing critical insights into resistance mechanisms and treatment efficacy prediction.

This study aims to evaluate the diagnostic performance (sensitivity, specificity, predictive values, accuracy) of 18F-FAPI-04 PET imaging in breast cancer. Additionally, it will monitor dynamic changes in FAP expression and tumor size during therapy, providing insights for patient stratification, clinical staging, treatment response assessment, early detection of resistance, and recurrence/metastasis, ultimately guiding personalized therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, any gender;
2. Clinically or pathologically confirmed diagnosis of breast cancer, or suspected recurrence/metastasis;
3. Presence of at least 1 measurable lesion (RECIST 1.1 criteria);
4. ECOG score 0-2 and expected survival ≥ 12 weeks;
5. Laboratory markers are met:

   Blood count: WBC ≥4.0×10⁹/L, PLT ≥100×10⁹/L, Hb ≥90 g/L Liver and kidney function: ALT/AST ≤ 2.5 × ULN, SCr ≤ 1.5 × ULN;
6. Signed informed consent.

Exclusion Criteria:

1. Major surgery or trauma within 4 weeks;
2. Severe infection, liver or kidney insufficiency;
3. History of allergies (developer components);
4. Pregnant/nursing female or not using effective contraception;
5. Inability to co-operate with PET (e.g. claustrophobia);
6. Any other situation that researchers considered it unsuitable to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to enroll 30 patients aged 18-75 years with clinically or pathologically confirmed breast cancer or suspected recurrence/metastasis, including both early-stage (I-II) and advanced-stage (III-IV) cases. The primary objective is to evaluate the diagnostic and therapeutic monitoring value of 18F-FAPI-04 PET for identifying primary tumors, metastatic lesions, and assessing treatment response. Exclusion criteria include: concurrent malignancies (except non-breast malignancies cured >5 years prior), severe hepatic or renal dysfunction, and pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
SUV | 2 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value (SUV) on PET

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No